CLINICAL TRIAL: NCT07098702
Title: Effectiveness of Ergonomic Practices on Quality of Breastfeeding Among Primiparous
Brief Title: Effect of Ergonomic Practices on Quality of Breastfeeding
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Aida Mohamed Ali Abd-Ellatif, Clinical Instructor at Technical Institute of Nursing, Faculty of Nursing, Mansoura University, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: effect of EP on QOB among pp
Record Dates: First submitted 2025-07-08; First posted 2025-08-01 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: we Search for the Effect of Ergonomic Practices on Quality of Breastfeeding
Keywords: Ergonomic Practices, Latch, Primiparous, Quality of Breastfeeding, Weight
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): In this group, the mothers will receive educational sessions regarding appropriate ergonomic practices during breastfeeding which include appropriate body mechanics, breastfeeding positions and breastfeeding pillows
  Interventions: Other: educational sessions and booklet
- control group (Experimental)
  Interventions: Other: No Interventions

INTERVENTIONS:
Other: educational sessions and booklet — educational sessions and booklet about ergonomic practices during breastfeeding which include appropriate body mechanics , breastfeeding positions, and use of breastfeeding pillows.
  Arms: intervention group
Other: No Interventions — In this group, the mothers will breastfeed their newborns according to the routine hospital postpartum instructions only.
  Arms: control group

SUMMARY:
This study aims to assess the effectiveness of ergonomic practices on quality of breastfeeding among primiparous.

DETAILED DESCRIPTION:
Prolonged discomfort experienced during lactation can significantly impede a mother's adjustment to the maternal role. This discomfort arises from suboptimal body positioning and extended periods of sitting during breastfeeding and some mothers stop breastfeeding as a result of that. Consequently, the promotion of maternal comfort during breastfeeding will enhance the quality of breastfeeding, and this will be achieved by encouraging mothers to assume appropriate body mechanics, appropriate breastfeeding positions, and use breastfeeding pillows during breastfeeding. Therefore, the researcher will conduct the current study.

ELIGIBILITY:
Inclusion Criteria:

* 1) Nulliparous women, 2) Mothers between the ages of 18 and 35, 3) Mothers who are in the third trimester, 4) Singleton pregnancy, 5) Mothers who have the intention of breastfeeding, and 6) Mothers who can read and write.

Exclusion Criteria:

* 1) Mothers with nipple problems, such as flat or inverted nipples, and 2) Mothers with medical or surgical problems interfering with breastfeeding.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — female pregnant mothers
Enrollment: 104 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
A LATCH score | At two weeks and two, four and six months after delivery
  A LATCH score of 0 to 3 is regarded as poor quality of breastfeeding, 4 to 7 is considered as moderate quality of breastfeeding, and 8 to 10 is considered as good quality of breastfeeding.

SECONDARY OUTCOMES:
Change in the growth chart of the infants | At two weeks and two, four, and six months after delivery
  neonates of the intervention group will exhibit better growth than neonates of the control group

CONTACTS AND LOCATIONS:
Overall Officials: Hanan El-Sayed Mohamed El-Sayed, Professor, Study Chair — Faculty of Nursing, Mansoura University, Egypt; Reda Abd El-Hady Ali Hemeda, Professor, Principal Investigator — Faculty of Medicine, Mansoura University, Egypt; Enas Sabry Fathy Elbeltagy, Lecturer, Principal Investigator — Faculty of Nursing, Mansoura University, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Efficacy of Counselling in Improving LATCH Score and Successful Breastfeeding: A Hospital-based Prospective Cohort Study. — https://doi.org/10.7860/JCDR/2022/56968.16685